CLINICAL TRIAL: NCT05443061
Title: Effect of Subcutaneous Nitroglycerin on the Prevention of Radial Artery Occlusion After Radial Artery Catheterization in Pediatric Patients - a Prospective Randomized Controlled Trial
Brief Title: Subcutaneous Nitroglycerin to Prevent Radial Artery Occlusion in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young-Eun Jang, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-2206-070-1332
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Arterial Line; Ischemia
Keywords: Radial Artery; Vascular Catheters
MeSH Terms: conditions — Ischemia | interventions — Nitroglycerin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitroglycerin (Experimental): Nitroglycerin 5mcg/kg (in 0.5cc) is subcutaneously injected before radial artery cannulation and before removal of the radial arterial catheter.
  Interventions: Drug: Nitroglycerin
- Control (Active Comparator): Normal saline (0.5cc) is subcutaneously injected before radial artery cannulation and before removal of the radial arterial catheter.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Nitroglycerin — Subcutaneous nitroglycerin injection to decrease the incidence of radial arterial occlusion after arterial catheter removal in pediatric patients.
  Arms: Nitroglycerin
Drug: Normal saline — Subcutaneous normal saline injection to decrease the incidence of radial arterial occlusion after arterial catheter removal in pediatric patients.
  Arms: Control

SUMMARY:
The primary objective of the study is to evaluate the vasodilative effect of subcutaneous nitroglycerin to prevent radial arterial occlusion(RAO) after removal of the radial arterial catheter in pediatric patients. The hypothesis of this study is that subcutaneous nitroglycerin will decrease the incidence of radial arterial occlusion after radial arterial catheter removal in pediatric patients by increasing the radial artery size. This is a single-center, double-blind, randomized, placebo-controlled study comparing the effect of subcutaneous nitroglycerin and saline on radial artery cannulation and catheter removal in pediatric patients. Prior to the procedure, each patient will be randomized into either the control arm, saline, or the study arm, nitroglycerin.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing General anesthesia
* Patients in the Intensive care unit
* Arterial cannulation for hemodynamic monitoring, or multiple blood sample

Exclusion Criteria:

* Unstable vital signs, significant arrhythmia or hypotension, Shock
* High risk of peripheral ischemia
* Skin disease, infection, hematoma, recent cannulation at the radial artery
* History of anaphylaxis to nitroglycerin

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
The incidence of radial arterial occlusion (RAO) (%) | After removal of the radial artery catheter (up to 24 hour)
  RAO is defined as no pulse oximeter wave at the index finger during compression of the ipsilateral ulnar artery.

SECONDARY OUTCOMES:
First attempt success rate (%) | During radial artery cannulation (up to 1 hour)
  Success at the first skin puncture
Size of radial artery (mm) | Before and after subcutaneous injection of drugs / Before and after catheterization / Before and after removal of the catheter (up to 1 hour)
  Internal diameter of radial artery
depth of radial artery (mm) | Before and after subcutaneous injection of drugs / Before and after catheterization / Before and after removal of the catheter (up to 1 hour)
  depth of radial artery from the skin
flow velocity of the radial artery (cm/s) | Before and after subcutaneous injection of drugs / Before and after catheterization / Before and after removal of the catheter (up to 1 hour)
  flow velocity of the radial artery measured by Doppler ultrasound
Perfusion index | Before and after subcutaneous injection of drugs / Before and after catheterization / Before and after removal of the catheter (up to 1 hour)
  Perfusion index measured by pulse oximeter sensor at the distally located index finger of radial arterial catheterization
Overall attempt (number) | During radial artery cannulation (up to 1 hour)
  Number of attempt of radial artery cannulation
Overall Procedure time (seconds) | During radial artery cannulation (up to 1 hour)
  From ultrasound guidance, to Arterial waveform
Overall success rate (%) | During radial artery cannulation (up to 1 hour)
  Success within 2 skin puncture and within 10 minutes
Incidence of posterior wall puncture (%) | During radial artery cannulation (up to 1 hour)
  Incidence of posterior wall (transfixation technique) puncture during radial arterial catherization
Number of arteries cannulated | During radial artery cannulation (up to 1 hour)
  Number of arteries cannulated for peripheral arterial catheterization
Malfunction of radial artery catheter | After radial artery cannulation assessed during anesthesia (per 24hour, up to 480 hour)
  Invasive blood pressure monitoring, Sampling (%)
Complication rate | After radial artery cannulation assessed up to PACU, PICU stay (per 24hour, up to 480 hour)
  Hematoma, Distal ischemia, Spasm accessed by ultrasound (%)
Duration of radial arterial catherization | After radial artery cannulation assessed during anesthesia (up to 480 hour)
  Duration of radial arterial catherization (hours, minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Eun Jang, MD, PhD, Principal Investigator — Clinical assistant professor, Department of anesthesiology and pain medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jang YE, Ji SH, Kim EH, Lee JH, Kim HS, Mossad EB, Kim JT. Subcutaneous Nitroglycerin for Radial Arterial Catheterization in Pediatric Patients: A Randomized Controlled Trial. Anesthesiology. 2020 Jul;133(1):53-63. doi: 10.1097/ALN.0000000000003308. PMID 32282432
- [Background] Jang YE, Cho SA, Ji SH, Kim EH, Lee JH, Kim HS, Kim JT. Smart Glasses for Radial Arterial Catheterization in Pediatric Patients: A Randomized Clinical Trial. Anesthesiology. 2021 Oct 1;135(4):612-620. doi: 10.1097/ALN.0000000000003914. PMID 34352073
- [Background] Jang YE, Kim EH, Lee JH, Kim HS, Kim JT. Guidewire-assisted vs. direct radial arterial cannulation in neonates and infants: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):738-744. doi: 10.1097/EJA.0000000000001064. PMID 31356376
- [Background] Kim EH, Lee JH, Song IK, Kim JT, Lee WJ, Kim HS. Posterior Tibial Artery as an Alternative to the Radial Artery for Arterial Cannulation Site in Small Children: A Randomized Controlled Study. Anesthesiology. 2017 Sep;127(3):423-431. doi: 10.1097/ALN.0000000000001774. PMID 28682811
- [Derived] Park JB, Ji SH, Kim EH, Lee JH, Kim HS, Kim JT, Jang YE. Subcutaneous Nitroglycerin to Prevent Radial Artery Occlusion in Pediatric Patients: A Randomized Clinical Trial. JAMA Pediatr. 2025 Dec 1;179(12):1283-1290. doi: 10.1001/jamapediatrics.2025.3652. PMID 41051743